CLINICAL TRIAL: NCT00006029
Title: A Phase I/II Study of Gemcitabine (GEMZAR)/Vinorelbine (NAVELBINE)/Liposomal Doxorubicin (DOXIL) in Relapsed/Refractory Hodgkin's Disease
Brief Title: Combination Chemotherapy in Treating Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-59804; CLB-59804; CDR0000068042 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence | interventions — Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vinorelbine + gemcitabine + doxorubicin - higher doses (Active Comparator): Patients who have not undergone prior transplantation receive vinorelbine, gemcitabine, and doxorubicin HCl liposome.
  Patients are followed every 6 months for 2 years and then annually for 6 years.
  Interventions: Drug: gemcitabine hydrochloride; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vinorelbine tartrate
- vinorelbine + gemcitabine + doxorubicin - lower doses (Experimental): Patients who have undergone prior transplantation receive lower doses of vinorelbine, gemcitabine, and doxorubicin HCl liposome.
  Patients are followed every 6 months for 2 years and then annually for 6 years.
  Interventions: Drug: gemcitabine hydrochloride; Drug: pegylated liposomal doxorubicin hydrochloride; Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: pegylated liposomal doxorubicin hydrochloride
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy in treating patients who have relapsed or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and toxicity of gemcitabine, vinorelbine, and doxorubicin HCl liposome in patients with relapsed or refractory Hodgkin's lymphoma.
* Determine the complete and partial response rates of patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study.

Phase I:

* Patients receive vinorelbine IV over 6-10 minutes, gemcitabine IV over 30 minutes, and doxorubicin HCl liposome IV over 30-60 minutes on days 1 and 8. Treatment continues every 21 days for 2-6 courses in the absence of unacceptable toxicity or disease progression. Patients who respond to treatment after 2 or more courses may stop protocol therapy to undergo peripheral blood stem cell transplantation.

Cohorts of 3-6 patients receive escalating doses of vinorelbine, gemcitabine, and doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive treatment with gemcitabine, vinorelbine, and doxorubicin HCl liposome at the recommended phase II dose.

Phase II:

* Patients are assigned to 1 of 2 treatment groups.

  * Group 1: Patients who have not undergone prior transplantation receive vinorelbine, gemcitabine, and doxorubicin HCl liposome as in phase I.
  * Group 2: Patients who have undergone prior transplantation receive lower doses of vinorelbine, gemcitabine, and doxorubicin HCl liposome as in group 1.

Patients are followed every 6 months for 2 years and then annually for 6 years.

PROJECTED ACCRUAL: Approximately 3-100 patients (3-42 for phase I and 20-58 for phase II [29 per group]) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma that is recurrent or refractory after standard chemotherapy

  * Core biopsy is acceptable if adequate tissue is obtained for primary diagnosis and immunophenotyping
  * Bone marrow biopsy is not acceptable as sole means of diagnosis
* Measurable disease

  * Tumor mass greater than 1 cm

PATIENT CHARACTERISTICS:

Age:

* Any age

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL unless history of Gilbert's disease
* AST no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* LVEF at least 45% by MUGA (for patients whose lifetime cumulative doxorubicin dose exceeds 400 mg/m^2)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior gemcitabine, vinorelbine, or doxorubicin HCl liposome
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormones except for nondisease-related conditions (e.g., insulin for diabetes) or steroids for adrenal failure
* No concurrent dexamethasone or other steroidal antiemetics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2000-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 4 years

SECONDARY OUTCOMES:
Overall survival | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L. Bartlett, MD, Study Chair — Washington University Siteman Cancer Center
Locations (76):
- United States (75):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Lai R, Bartlett NL, Mackey JR, Jung SH, Johnson JL, Cook JR, Jones D, Cass CE, Young JD, Said J, Cheson B, Hsi ED. High expression of nucleoside transporter protein hENT1 in Reed-Sternberg cells is associated with treatment failure in relapsed/refractory Hodgkin lymphoma patients treated with gemcitabine, vinorelbine and liposomal doxorubicin - a CALGB 59804 correlative study. Leuk Lymphoma. 2008 Jun;49(6):1202-5. doi: 10.1080/10428190802094237. No abstract available. PMID 18452103
- [Result] Bartlett NL, Niedzwiecki D, Johnson JL, Friedberg JW, Johnson KB, van Besien K, Zelenetz AD, Cheson BD, Canellos GP; Cancer Leukemia Group B. Gemcitabine, vinorelbine, and pegylated liposomal doxorubicin (GVD), a salvage regimen in relapsed Hodgkin's lymphoma: CALGB 59804. Ann Oncol. 2007 Jun;18(6):1071-9. doi: 10.1093/annonc/mdm090. Epub 2007 Apr 10. PMID 17426059
- [Result] Bartlett N, Niedzwiecki D, Johnson J, et al.: A phase I/II study of gemcitabine, vinorelbine, and liposomal doxorubicin for relapsed Hodgkin's disease: preliminary results of CALGB 59804. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2275, 566, 2003.